CLINICAL TRIAL: NCT04680793
Title: Effects of a Multidisciplinary Outpatient Rehabilitation Program on Physical Capacity and Quality of Life in Patients With Ehlers-Danlos Syndrome.
Brief Title: Effects of a Multidisciplinary Outpatient Rehabilitation Program in Patients With Ehlers-Danlos Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hakimi Adrien (Other)
Responsible Party: Sponsor-Investigator, Hakimi Adrien, PhD Student, Clinique de la Mitterie
Organization: Clinique de la Mitterie (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A02154-53
Record Dates: First submitted 2020-12-16; First posted 2020-12-23 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Ehlers-Danlos Syndrome
Keywords: Rehabilitation; Ehlers-Danlos syndrome; Quality of life; Physical capacity
MeSH Terms: conditions — Ehlers-Danlos Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Patients are assessed 9 weeks before the start of the program, at the beginning and at the end of the program, and 6 weeks and 6 months after the end of the program. The 9-week period before the program is used as a control condition. It is of the same duration as the program, which also lasts 9 weeks. Patients are asked not to change their lifestyle during the 9-week period before the rehabilitation program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EDS Patients (Other): No intervention during the control period (9 weeks) and then experimental during the rehabilitation stage (9 weeks).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The program takes place over a total period of 9 weeks: for 4 weeks they will be cared for two days a week, then after a week's break, for 4 weeks they will be cared for three days a week for a total of approximately 80 hours of care. The program is multidisciplinary and includes: balneotherapy, ergometry, occupational therapy, gymnastics, physiotherapy, walking, sophrology, yoga as well as different workshops for the therapeutic education of the patient led by several professionals (dieticians, physiotherapists, doctors, psychologists).

SUMMARY:
The management of patients with Ehlers-Danlos syndrome (EDS) is still underdeveloped in healthcare institutions in France. Although multidisciplinary management through exercise rehabilitation has demonstrated its benefits in many chronic pathologies, it has not been evaluated for EDS. As a result, to date there is no evidence of its effectiveness in patients with EDS. The objective of this study is therefore to objectively evaluate the effectiveness of such a treatment on the different dimensions of these patients' health.

ELIGIBILITY:
Inclusion Criteria:

* EDS diagnosis.
* Inclusion in the rehabilitation program.

Exclusion Criteria:

* Absolute and relative cardio-vascular contraindications to rehabilitation.
* Other contraindications to exercise.
* Psychological contraindication (Beck questionnaire score ≥ 20)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Distance covered in the 6-minute walk test | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months

SECONDARY OUTCOMES:
Other data from the 6-minute walk test | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months
Time of an endurance test on a cyclo-ergometer | Baseline ; 9 weeks
Area swept by the gravity center during a balance test on a posturological platform | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months
  Four balance tests : bipodal with eyes open, bipodal with eyes closed and unipodal with eyes open on the two sides
Tampa scale for kinesiophobia (questionnaire) | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months
Brief pain inventory (questionnaire) | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months
Nijmegen questionnaire | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months
Multidimensional fatigue inventory (questionnaire) | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months
Medical outcome study short form 36 (questionnaire) | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months
Hospital anxiety and depression scale (questionnaire) | 9 weeks before baseline ; Baseline ; 9 weeks ; 15 weeks ; 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MUCCI, Prof., Study Director — URePSSS; Cyrille BERGOIN, Dr., Principal Investigator — Clinique de la Mitterie
Locations (1):
- Clinique de la Mitterie, Lomme, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hakimi A, Bergoin C, De Jesus A, Hoorelbeke A, Ramon P, Florea O, Fabre C, Mucci P. Multiple Sustainable Benefits of a Rehabilitation Program in Therapeutic Management of Hypermobile Ehlers-Danlos Syndrome: A Prospective and Controlled Study at Short- and Medium-Term. Arch Phys Med Rehabil. 2023 Dec;104(12):2059-2066. doi: 10.1016/j.apmr.2023.06.012. Epub 2023 Jul 4. PMID 37406924
- [Derived] Hakimi A, Bergoin C, Mucci P. Evidence of ventilatory constraints during exercise in hypermobile Ehlers-Danlos syndrome. Eur J Appl Physiol. 2022 Nov;122(11):2367-2374. doi: 10.1007/s00421-022-05017-y. Epub 2022 Aug 8. PMID 35941284